CLINICAL TRIAL: NCT00074516
Title: Renal Transplantation in Recipients With Nephropathic Cystinosis
Brief Title: Kidney Transplantation in Patients With Cystinosis
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040057; 04-DK-0057
Record Dates: First submitted 2003-12-12; First posted 2003-12-15 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2014-06-11

CONDITIONS: Cystinosis
Keywords: Immunosuppression; Kidney; Cysteamine; Steroid-Free; Outcomes
MeSH Terms: conditions — Cystinosis

SUMMARY:
This study will test the effectiveness of a combination of anti-rejection medicines in preventing complications typically seen in cystinosis patients undergoing kidney transplants. Cystinosis is a rare disease affecting children that causes growth retardation and kidney failure. Kidney transplant is the standard treatment for kidney failure in these patients, followed by immunosuppression to prevent organ rejection. The standard drug regimen for immunosuppression includes steroids, which can lead to other serious complications. This study will look at combination therapy that does not include steroids.

Patients 7 years of age and older with cystinosis who are candidates for a kidney transplant at the National Institutes of Health Clinical Center may be eligible for this 5-year study. Candidates will be screened with a medical history, physical examination, and blood tests.

Participants will undergo the following tests and procedures:

1. Kidney transplant: Patients undergo kidney transplant surgery under general anesthesia.
2. Central line placement: A large intravenous catheter (plastic tube, or IV line) is placed in a vein in the chest or neck under local anesthesia before the transplant surgery. The line remains in place for some time during the hospitalization to administer immunosuppressive medications, antibiotics, and blood, if needed. The line is also used to collect blood samples.
3. Leukapheresis: This procedure for collecting white blood cells is done before the transplant. The cells are studied to evaluate the patient's immune system. Whole blood is withdrawn through a catheter in an arm vein or through the central line and directed into a machine that separates the blood components by spinning. The white cells are removed and the red cells and plasma are returned to the body.
4. Immunosuppressive medication following transplantation

   * Adults receive thymoglobulin at the time of the transplant and for 3 days after surgery; mycophenolate mofetil daily after the transplant; tacrolimus twice a day once the kidney is working well; and sirolimus daily.
   * Children receive daclizumab the day of the transplant, day 4 after surgery, and at weeks 2, 4, 6, 8, 11, 15, 19, and 23, and mycophenolate mofetil daily after the transplant.
5. Follow-up visits: After discharge from the hospital, patients return to the Clinical Center for follow-up at 6 months, at 1 year, and then yearly for 5 years. A physical examination is done the first four visits, and blood and urine samples are collected at every visit. Kidney biopsies (removal of a small amount of kidney tissue through a thin needle) are done at 6 months, 1, 3, and 5 years after the transplant. The biopsied tissue is examined to evaluate how well the kidney is responding to the immunosuppression medicines, to determine whether more or less medication is needed, and to evaluate how the patient is responding to the donor kidney.
6. Routine laboratory tests, coordinated by the patient's local physician, are done 2 to 3 times a week for the first 2 to 3 months after transplantation, then weekly for several more months, and at least monthly for life.

DETAILED DESCRIPTION:
Cystinosis is an autosomal recessive disorder due to impaired cystine transport across the lysosomal membrane, resulting in abnormal cystine accumulation throughout the body. Fanconi syndrome manifests in the first year of life, and end-stage renal failure occurs at ~10 years of age, requiring dialysis or kidney transplantation. Oral cysteamine therapy delays but does not always prevent the need for a renal allograft in cystinosis, which accounts for ~3% of all pediatric transplants in the United States. With improvements in immunosuppression, short-term graft and patient survival is quite good for cystinosis patients, although not as good as for patients with ESRD due to structural defects. Long-term graft survival can be affected by the non-renal complications of cystinosis, which persist after renal transplantation.

The aim of this study is to establish standards for the transplantation of kidneys into patients with nephropathic cystinosis using steroid-sparing immunosuppression. Our goals are to:

1. Analyze the long and short term outcome of cystinosis patients following living and cadaveric kidney transplantation using steroid-free immunosuppression;
2. Determine a consistent clinical approach to recipients with cystinosis in the immediate post-operative period, specifically regarding fluid and electrolyte management, retention of native kidneys, and timing of the re-initiation of cystinosis therapy after transplantation;
3. Assess the immunologic impact of cystinosis by monitoring immune responses using a number of in vitro assays.

In this study, patients will receive a living donor or cadaveric kidney transplant with steroid free immunosuppression. Graft function, histology and graft and patient survival will be measured. Progression of cystinosis in other organ systems will be monitored. Additional studies on the graft will include transcriptional analysis of inflammatory and immunologic mediators. Serum will be assayed for inflammatory mediators and peripheral white blood cells assayed for immune function. This study will represent the first comprehensive, prospective analysis of kidney transplantation in patients with cystinosis.

ELIGIBILITY:
* INCLUSION CRITERIA:

Candidates for a kidney transplant at the National Institutes of Health Clinical Center.

Ability and willingness to provide informed consent (adults greater than or equal to 18.0 years) or assent (children greater than or equal to 7 years and less than 18.0 years).

Willingness to travel to the Clinical Center for protocol samples to be collected and the ability to send samples from a local collection source and mail them overnight.

EXCLUSION CRITERIA:

Inability or unwillingness to comply with protocol, or to provide informed consent. Criteria include a history of noncompliance, circumstances where compliance with protocol requirements is not feasible due to living conditions, travel restrictions, lack of access to urgent medical services, or access to anti-rejection drugs once the study is completed.

Any active malignancy or history of a hematogenous malignancy or lymphoma. Patients with primary, cutaneous basal cell or squamous cell cancers may be enrolled providing the lesions are appropriately treated prior to transplantation.

Significant coagulopathy or requirement for anticoagulation therapy that would contraindicate allograft biopsy.

Any known immunodeficiency syndrome.

Peak panel reactive antibody greater than 20% or historically positive crossmatch due to HLA-specific antibodies.

Prior kidney graft survival less than 3 years or positive T or B cell crossmatch in patients receiving repeat kidney allograft.

Historical or current positive T cell cross match between donor and recipient.

Pregnancy or unwillingness to practice an approved method of birth control. Acceptable methods of birth control may include barrier methods, oral contraceptives, Norplant, Depo-Provera, or partner sterility.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2003-12-10; Study Completion 2014-06-11

CONTACTS AND LOCATIONS:
Overall Officials: Monique E Cho, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gahl WA, Bashan N, Tietze F, Bernardini I, Schulman JD. Cystine transport is defective in isolated leukocyte lysosomes from patients with cystinosis. Science. 1982 Sep 24;217(4566):1263-5. doi: 10.1126/science.7112129.
- [Background] Town M, Jean G, Cherqui S, Attard M, Forestier L, Whitmore SA, Callen DF, Gribouval O, Broyer M, Bates GP, van't Hoff W, Antignac C. A novel gene encoding an integral membrane protein is mutated in nephropathic cystinosis. Nat Genet. 1998 Apr;18(4):319-24. doi: 10.1038/ng0498-319. PMID 9537412
- [Background] Gahl WA, Thoene JG, Schneider JA. Cystinosis. N Engl J Med. 2002 Jul 11;347(2):111-21. doi: 10.1056/NEJMra020552. No abstract available. PMID 12110740